CLINICAL TRIAL: NCT01640431
Title: Lumbar Segmental Stabilization and TENS in Lumbar Disc Herniation: a Randomized Clinical Trial
Brief Title: Lumbar Segmental Stabilization and TENS in Lumbar Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fisio2011
Record Dates: First submitted 2012-07-03; First posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Lumbar Spine Disc Herniation
Keywords: lumbar disc herniation; clinical trial; exercise therapy; TENS
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lumbar stabilization exercises (Experimental): In the Segmental Stabilization group exercises the focus is on the transversus abdominis and lumbar multifidus muscles.
  Interventions: Other: Lumbar stabilization exercises
- TENS group (Experimental): In this group, patients are treated with TENS in the lumbar region for an hour.
  Interventions: Other: Lumbar stabilization exercises

INTERVENTIONS:
Other: Lumbar stabilization exercises — The patients performed exercises for the transversus abdominis and lumbar multifidus muscles for an hour twice a week.

SUMMARY:
The purpose of this study was to compare the efficacy of method Lumbar Segmental Stabilization and transcutaneous electrical nerve stimulation (TENS) on pain, functional disability and ability to activate the transversus abdominis (TrA) of individuals with chronic back pain caused by disc herniation.

DETAILED DESCRIPTION:
Objective: To contrast the efficacy efficacy of method Lumbar Segmental Stabilization and TENS on pain, functional capacity and ability to activate the TrA of individuals with chronic back pain caused by disc herniation.

Design: Sixty patients are being randomized into two groups namely: Lumbar Segmental Stabilization (LS ) (specific exercises for the muscles transversus abdominis and lumbar multifidus) (n = 30) and TENS group (TG) (n = 30) receiving assistance under a current of transcutaneous electrical nerve stimulation (TENS). Groups were contrasted regarding pain (visual analogical scale and McGill pain questionnaire), functional disability (Oswestry disability questionnaire) and TrA muscle activation capacity (Pressure Biofeedback Unit = PBU). The program lasts for 8 weeks, and sessions happen twice a week, with duration of one hour each. Evaluations will be performed before, after and with a follow-up six months after treatment. Significance level is established at 5%.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain (pain for more than three months) or sciatica caused by disc herniation diagnosed by magnetic resonance imaging or computed tomography

Exclusion Criteria:

* prior back surgery,
* cancer,
* rheumatic diseases or infection.

Patients involved in sports or resistance training for the lumbar spine during the three months prior to the beginning of treatment or other causes of pain and sciatica such as lumbar spinal canal stenosis and lumbar spondylolisthesis have also been excluded.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Pain. | 8 weeks
  The pain will be assessed with the visual analogical scale and McGill pain questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio R França, MsC, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rackwitz B, de Bie R, Limm H, von Garnier K, Ewert T, Stucki G. Segmental stabilizing exercises and low back pain. What is the evidence? A systematic review of randomized controlled trials. Clin Rehabil. 2006 Jul;20(7):553-67. doi: 10.1191/0269215506cr977oa. PMID 16894798
- [Derived] Franca FJR, Callegari B, Ramos LAV, Burke TN, Magalhaes MO, Comachio J, CarvalhoSilva APMC, Almeida GPL, Marques AP. Motor Control Training Compared With Transcutaneous Electrical Nerve Stimulation in Patients With Disc Herniation With Associated Radiculopathy: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2019 Mar;98(3):207-214. doi: 10.1097/PHM.0000000000001048. PMID 30247159